CLINICAL TRIAL: NCT05342675
Title: Effect of Post-Procedural Rapid Rollover on Pneumothorax After Percutaneous CT-Guided Lung Biopsy: A Randomized Controlled Trial
Brief Title: Effect of Rapid Rollover on Pneumothorax After CT-Guided Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-36288
Record Dates: First submitted 2022-04-01; First posted 2022-04-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Pneumothorax
Keywords: CT-guided lung biopsy; Chest tube
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Eligible patients will be randomized into either the control group (standard protocol CT-guided lung biopsy) or the rapid rollover group (immediate reposition with biopsy site down).
Who Masked: Investigator
Masking Description: Interpreting radiologists of the post-biopsy CTs and radiographs will be blinded to whether the patient is in the control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Rollover (Experimental): Participants will have their body re-positioned upon being transferred to the stretcher from the CT scanner table such that the biopsy site is down. Participants will be maintained in the same position for the post-biopsy CT scanner as well as in the post-procedure recovery area for a minimum of 2 hours.
  Interventions: Procedure: Rapid Rollover
- Control (No Intervention): CT-guided lung biopsy will be performed per standard protocols

INTERVENTIONS:
Procedure: Rapid Rollover — Repositioning of the participant post biopsy
  Arms: Rapid Rollover

SUMMARY:
Pneumothorax is the most common complication after CT-guided lung biopsy, and several techniques have been proposed to reduce the risk. Among them, rapid rollover is the maneuver to immediately reposition the patient, with biopsy-side down after removal of biopsy needle. It has been theorized that the technique reduces the size of alveoli surrounding the needle tract, leading to airway closure and reduction in the alveolar-to-pleural pressure gradient, thereby preventing pneumothorax. The aim of this study is to evaluate the effectiveness of rapid rollover in reducing the risk of radiographically detectable pneumothorax and the rate of chest tube insertion.

Patients undergoing CT-guided lung biopsy for any indication will be recruited and randomized into either rapid rollover group or control group. In the control group, CT guided lung biopsy will be performed per standard protocols; in the rapid rollover group, the biopsy will also be performed per the same protocol with the addition of rapid rollover at the end of the procedure. For both groups, the primary outcome would be new or enlarging pneumothorax detected on post-biopsy radiographs, and the secondary outcome would be the risk of pneumothorax necessitating chest tube insertion, all complications associated with CT guided lung biopsy, time to complication development, and patient experience in each arm.

DETAILED DESCRIPTION:
All patients will undergo CT-guided lung biopsy by the best approach decided by the primary operator. Randomization will be performed based on parity of patients' medical record numbers, which were assigned randomly at their first presentation. Patients with even medical record numbers will be assigned to the control group and patients with odd medical record number will be assigned to the intervention group.

In the rapid rollover group, patients will be repositioned upon being transferred from the CT scanner table to the stretcher such that the biopsy site is down. Patient in the intervention arm will be maintained in the same position in the post-procedure recovery area for at least 2 hours if patients can tolerate. Anyone who maintains the biopsy-site down position for at least 30 minutes after repositioning in the intervention group will be considered as completion of the intervention. Patients who are in the controlled arm may choose the most comfortable position per their preferences. All patients will be monitored for at least 2 hours, after which a 0-1 hour optional post-biopsy radiograph and 2-hour follow-up radiograph will be obtained to assess for pneumothorax per the standard current protocol. Further follow-up radiograph may be obtained if the patient did not receive the 0-1 hour radiograph and the 2-hour radiograph was positive for pneumothorax that is not large enough to require immediate chest tube insertion. Interpreting radiologists of the post-biopsy radiographs will be blinded to whether the patient is in the control or intervention group.

A survey will be given to the patients in post-anesthesia care unit by nurses before they are discharged.

Multiple patient-, lesion- and technique-specific factors will be recorded:

Patient-specific factors:

* Age
* Gender
* Indication of lung biopsy
* History of underlying lung disease
* History of tobacco use
* Prior lung surgery or radiation

Lesion-specific factors:

* Location
* Size
* Morphology
* Shortest distance from pleura Technique-specific factors
* Approach
* Patient positioning during procedure
* Number of times crossing the pleura
* Number of times crossing the fissure
* Number of fine needle aspirations (FNAs)
* Number of core biopsies
* Needle-path length
* Needle-pleura angle
* Co-axial size
* Duration of biopsy site down time and number of turns as tolerated by the patient
* Use of blood patch

ELIGIBILITY:
Inclusion Criteria:

* All patients who are referred to the Department of Radiology and Biomedical Imaging Cardiac and Pulmonary Imaging section for CT-guided lung biopsy will be screened for eligibility. All eligible patients will be enrolled. Patients who develop intra-procedural pneumothorax will be analyzed but excluded from the final analysis.

Exclusion Criteria:

* Patients with chest wall, subpleural or mediastinal lesions
* Patients who develop intra-procedural pneumothorax
* Patients who are biopsied by a prone approach
* Patients who are repositioned intra-procedurally
* Patients who are unable to tolerate reposition or have spinal precautions
* Patients who develop hemothorax and a chest tube is inserted for this indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Radiographically detectable pneumothorax | 2 hours after biopsy
  New or enlarging pneumothorax (from intraprocedural CT) which is detectable on post biopsy radiograph. The size of the pneumothorax will be measured in terms of the distance between visceral and parietal pleura. The severity of pneumothorax will be assessed using CTCAE 5.0.

SECONDARY OUTCOMES:
Chest tube insertion | 24 hours for overnight observation
  Pneumothorax that requires chest tube insertion or other operative interventions (or CTCAE 5.0 grade 2 and above). While the decision to intervene could be operator-dependent, chest tube insertion takes place at our institution for patients with 1) enlarging or symptomatic small pneumothorax, and 2) moderate pneumothorax regardless of symptoms.
Enlarging pneumothorax | From 2 hours post biopsy to patient being discharged home.
  Enlarging pneumothorax from baseline pneumothorax > 3 mm (distance between visceral and parietal pleura measured on chest radiograph) accounting for redistribution of air and projection.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Sohn, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
Study results will be published.

REFERENCES:
- [Background] Hiraki T, Mimura H, Gobara H, Shibamoto K, Inoue D, Matsui Y, Kanazawa S. Incidence of and risk factors for pneumothorax and chest tube placement after CT fluoroscopy-guided percutaneous lung biopsy: retrospective analysis of the procedures conducted over a 9-year period. AJR Am J Roentgenol. 2010 Mar;194(3):809-14. doi: 10.2214/AJR.09.3224. PMID 20173164
- [Background] Kim JI, Park CM, Lee SM, Goo JM. Rapid needle-out patient-rollover approach after cone beam CT-guided lung biopsy: effect on pneumothorax rate in 1,191 consecutive patients. Eur Radiol. 2015 Jul;25(7):1845-53. doi: 10.1007/s00330-015-3601-y. Epub 2015 Feb 1. PMID 25636421
- [Background] O'Neill AC, McCarthy C, Ridge CA, Mitchell P, Hanrahan E, Butler M, Keane MP, Dodd JD. Rapid needle-out patient-rollover time after percutaneous CT-guided transthoracic biopsy of lung nodules: effect on pneumothorax rate. Radiology. 2012 Jan;262(1):314-9. doi: 10.1148/radiol.11103506. Epub 2011 Nov 21. PMID 22106349
- [Background] Najafi A, Al Ahmar M, Bonnet B, Delpla A, Kobe A, Madani K, Roux C, Deschamps F, de Baere T, Tselikas L. The PEARL Approach for CT-guided Lung Biopsy: Assessment of Complication Rate. Radiology. 2022 Feb;302(2):473-480. doi: 10.1148/radiol.2021210360. Epub 2021 Nov 2. PMID 34726537
- [Background] Tanisaro K. Patient positioning after fine needle lung biopsy-effect on pneumothorax rate. Acta Radiol. 2003 Jan;44(1):52-5. PMID 12630999
- [Background] Collings CL, Westcott JL, Banson NL, Lange RC. Pneumothorax and dependent versus nondependent patient position after needle biopsy of the lung. Radiology. 1999 Jan;210(1):59-64. doi: 10.1148/radiology.210.1.r99ja1759. PMID 9885587
- [Background] Heerink WJ, de Bock GH, de Jonge GJ, Groen HJ, Vliegenthart R, Oudkerk M. Complication rates of CT-guided transthoracic lung biopsy: meta-analysis. Eur Radiol. 2017 Jan;27(1):138-148. doi: 10.1007/s00330-016-4357-8. Epub 2016 Apr 23. PMID 27108299
- [Background] Huo YR, Chan MV, Habib AR, Lui I, Ridley L. Pneumothorax rates in CT-Guided lung biopsies: a comprehensive systematic review and meta-analysis of risk factors. Br J Radiol. 2020 Apr 1;93(1108):20190866. doi: 10.1259/bjr.20190866. Epub 2020 Jan 3. PMID 31860329
- [Background] Huo YR, Chan MV, Habib AR, Lui I, Ridley L. Post-Biopsy Manoeuvres to Reduce Pneumothorax Incidence in CT-Guided Transthoracic Lung Biopsies: A Systematic Review and Meta-analysis. Cardiovasc Intervent Radiol. 2019 Aug;42(8):1062-1072. doi: 10.1007/s00270-019-02196-8. Epub 2019 Mar 12. PMID 30863965
- [Background] Tomiyama N, Yasuhara Y, Nakajima Y, Adachi S, Arai Y, Kusumoto M, Eguchi K, Kuriyama K, Sakai F, Noguchi M, Murata K, Murayama S, Mochizuki T, Mori K, Yamada K. CT-guided needle biopsy of lung lesions: a survey of severe complication based on 9783 biopsies in Japan. Eur J Radiol. 2006 Jul;59(1):60-4. doi: 10.1016/j.ejrad.2006.02.001. Epub 2006 Mar 10. PMID 16530369